CLINICAL TRIAL: NCT07050017
Title: High Milk Protein Content Reduces ad Libitum Post-exercise Energy Intake Without Altering Appetite in Active Males
Brief Title: Impact of Protein Content of Milk on Post-Exercise Appetite and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Tunçil, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SBF-25-059
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Appetite; Energy Intake; Post-exercise; Negative Energy Balance
Keywords: milk; high-protein milk; protein; post-exercise; appetite; energy intake

STUDY DESIGN:
Intervention Model Description: All participants will attend 5 visits. Two of them are pre-screening visits.
Who Masked: Participant, Care Provider
Masking Description: The beverages will be administered in opaque bottles in a randomized order. Both the participants and the researchers will remain blinded to the content of the beverages until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- carbohydrate control drink: isoenergetic and isovolumetric with milk beverages. (Active Comparator): Isoenergetic and isovolumetric with milk beverages
  Interventions: Behavioral: The study will investigate how different amounts of protein (0 g, 15 g, and 30 g) in post-exercise beverages affect appetite and energy intake following endurance exercise.
- regular milk (Experimental): containing 15 g protein
  Interventions: Behavioral: The study will investigate how different amounts of protein (0 g, 15 g, and 30 g) in post-exercise beverages affect appetite and energy intake following endurance exercise.
- high-protein milk (Experimental): containing 30 g protein
  Interventions: Behavioral: The study will investigate how different amounts of protein (0 g, 15 g, and 30 g) in post-exercise beverages affect appetite and energy intake following endurance exercise.

INTERVENTIONS:
Behavioral: The study will investigate how different amounts of protein (0 g, 15 g, and 30 g) in post-exercise beverages affect appetite and energy intake following endurance exercise. — The study will investigate how different amounts of protein (carbohydrate control drink : 0 g, reguler milk : 15 g, and high-protein milk : 30 g) in post-exercise beverages affect appetite and energy intake following endurance exercise.

SUMMARY:
This study aims to investigate the acute effects of consuming milk beverages with different protein content on subjective appetite and energy intake in healthy adults following endurance exercise. Participants will complete an endurance exercise protocol and then consume one of three beverages: a high-protein milk, a regular-protein milk, or an isoenergetic and isovolumetric carbohydrate control drink. Subjective appetite ratings will be assessed using visual analogue scales (VAS) at multiple time points after beverage consumption. Appetite-related hormonal responses, including insulin and acylated ghrelin, will be measured via blood samples. Energy intake will be assessed through an ad libitum test meal. This study will help determine whether different types of milk consumed post-exercise influence appetite regulation, hormonal response, and subsequent energy intake.

DETAILED DESCRIPTION:
The primary objective of this randomized, double-blind, crossover clinical trial is to evaluate the acute effects of post-endurance exercise consumption of milk beverages with varying protein content on subjective appetite, circulating appetite-related hormones, and subsequent ad libitum energy intake in healthy, recreationally active adult males. The study will recruit at least 12 healthy male participants aged 18-39 years who have been regularly engaged in endurance-based physical activity (e.g., cycling, running, triathlon, orienteering, team sports) for a minimum of one year, with a training frequency of at least three sessions per week lasting 60-90 minutes each. Participants will complete five laboratory visits under a crossover design with a minimum one-week washout period between intervention conditions. The first two sessions will consist of pre-study visits (screening, anthropometric assessments, VO₂max testing, and familiarization). The remaining three visits will involve the ingestion of one of the following beverages in a randomized order: standard-protein milk (0 g protein), high-protein milk (30 g protein), or an isoenergetic carbohydrate-based control beverage (0 g protein). All beverages will be isocaloric and isovolumetric and provided in opaque bottles to ensure double-blind conditions. On each intervention day, participants will perform a steady-state endurance exercise protocol using a calibrated cycle ergometer, followed immediately by the ingestion of one of the test beverages. Appetite will be assessed subjectively using validated Visual Analogue Scales (VAS) at predefined intervals. Venous blood samples will be collected to analyze concentrations of insulin and acylated ghrelin as objective biomarkers of appetite regulation. One hour after beverage consumption, an ad libitum test meal will be provided to quantify subsequent energy intake. The total caloric intake and macronutrient distribution will be recorded and analyzed. This study is designed to provide insight into the role of post-exercise milk consumption-specifically the influence of protein content-on short-term appetite modulation and energy intake regulation in recreationally trained individuals.

ELIGIBILITY:
Inclusion Criteria:

* The study will include healthy, physically active male participants aged 18-39 years who have been engaging in recreational endurance sports (such as cycling, running, triathlon, orienteering, or team sports) for at least one year, with a minimum frequency of 3 sessions per week lasting 60-90 minutes.

Exclusion Criteria:

* Current smoker
* Chronic or excessive alcohol consumption
* Use of supplements and/or chronic medications that may affect appetite
* Presence of cardiac, hepatic, renal, pulmonary, neurological, hematological, gastrointestinal, diabetic, thyroid, or psychiatric disorders, and/or musculoskeletal conditions that may limit exercise participation
* Allergy or intolerance to any of the foods or beverages to be consumed during the study
* Unstable body weight (e.g., weight loss greater than 1 kg in the past week)
* Currently following a weight-loss diet
* Diagnosed eating disorders or individuals who cognitively restrict food intake (to be assessed using the Three-Factor Eating Questionnaire)

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
energy intake | From enrollment to the end of treatment at 3 weeks.
  Energy intake will be measured through an ad libitum meal provided after the exercise.

SECONDARY OUTCOMES:
acylated ghrelin (pg/mL) | From enrollment to the end of treatment at 3 weeks.
  Plasma acyl ghrelin will be measured as an indicator of appetite.
Insulin (pmol/L) | From enrollment to the end of treatment at 3 weeks.
  Plasma insulin will be measured as an indicator of appetite and glucose metabolism.
subjective appetite | From enrollment to the end of treatment at 3 weeks.
  Subjective appetite will be assessed using Visual Analogue Scales (mm).

CONTACTS AND LOCATIONS:
Overall Officials: muhammed atakan, Associate Professor, Study Chair — Hacettepe University; zeynep ergün, PHD student, Study Chair — Hacettepe University; süleyman bulut, Associate Professor, Study Chair — Hacettepe University; hüsrev turnagöl, professor, Study Chair — Hacettepe University; tahir hazır, professor, Study Chair — Hacettepe University; yiğitcan karanfil, Assistant professor, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No